CLINICAL TRIAL: NCT01025856
Title: Combined Nutritional and Exercise Strategies to Reduce Liver Fat Content in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, PA, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46/09
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Postprandial Lipids Metabolism; Type 2 Diabetes
Keywords: liver fat; postprandial lipids metabolism; diet; exercise; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- high fibre/low glycemic index diet - P A (Active Comparator): patients will follow for two months a diet high fibre/low glycemic index without physical activity program
  Interventions: Other: High fibre/low glycemic index diet-PA
- Rich in MUFA diet - PA (Active Comparator): Patients will follow for two months a rich in MUFA diet without a physical activity program.
  Interventions: Other: Rich in MUFA diet -PA
- high fibre/low glycemic index diet+PA (Active Comparator): Patients will follow for two months a high fibre and low glycemic index diet associated with a physical activity program.
  Interventions: Other: high fiber/low glycemic index diet + pa
- Rich in MUFA diet+PA (Active Comparator): Patients will follow for 2 months a rich in MUFA diet with a physical activity program.
  Interventions: Other: Rich in MUFA diet+PA

INTERVENTIONS:
Other: Rich in MUFA diet -PA — The patients will follow a rich in MUFA diet without a physical activity program.
  Arms: Rich in MUFA diet - PA
Other: high fiber/low glycemic index diet + pa — patients will follow for two months a high fibre/ low glycemic index diet with a physical activity program.
  Arms: high fibre/low glycemic index diet+PA
Other: Rich in MUFA diet+PA — Patients will follow for two months a rich in MUFA diet with a physical activity program.
  Arms: Rich in MUFA diet+PA
Other: High fibre/low glycemic index diet-PA — Patients will follow for two months a high fibre/low glycemic index diet without a physical activity program.
  Arms: high fibre/low glycemic index diet - P A

SUMMARY:
The aim of this study will be to evaluate in patients with type 2 diabetes the effects on liver fat of an intervention with a diet relatively rich in CHO/rich in fibre/low GI or a diet rich in MUFA, either combined or not with a structured program of physical exercise, with emphasis on mechanisms possibly underlining these effects, namely changes in postprandial triglyceride-rich lipoproteins, body fat distribution, insulin sensitivity, oxidative stress and inflammation, adipose tissue lipolytic activities, aerobic capacity and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women
* Age 35-65 years
* BMI 27- 34 kg/m2
* HbA1c <8%
* Fasting plasma cholesterol <250 mg/dl
* Fasting plasma triglycerides <300 mg/dl

Exclusion Criteria:

* Hypolipidemic drugs
* Plasma creatinine >1.7 mg/dl transaminases > 2 norma values
* Ischemic heart disease or positive treadmill stress test
* High intensity regular physical activity
* Any disease or chronic or/and acute condition contraindicating physical activity(anaemia, and infectious, neoplastic, neurological and osteoarticular diseases).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Liver fat content | 0 and 8 weeks
postprandial lipids metabolism | 0 and 8 weeks

SECONDARY OUTCOMES:
changes in body fat distribution | 0 and 8 weeks
oxidative stress and inflammation | 0 and 8 weeks
adipose tissue lipolytic activities | 0 and 8 weeks

REFERENCES:
- [Derived] Bozzetto L, Costabile G, Luongo D, Naviglio D, Cicala V, Piantadosi C, Patti L, Cipriano P, Annuzzi G, Rivellese AA. Reduction in liver fat by dietary MUFA in type 2 diabetes is helped by enhanced hepatic fat oxidation. Diabetologia. 2016 Dec;59(12):2697-2701. doi: 10.1007/s00125-016-4110-5. Epub 2016 Sep 20. PMID 27650287
- [Derived] Bozzetto L, Annuzzi G, Costabile G, Costagliola L, Giorgini M, Alderisio A, Strazzullo A, Patti L, Cipriano P, Mangione A, Vitelli A, Vigorito C, Riccardi G, Rivellese AA. A CHO/fibre diet reduces and a MUFA diet increases postprandial lipaemia in type 2 diabetes: no supplementary effects of low-volume physical training. Acta Diabetol. 2014;51(3):385-93. doi: 10.1007/s00592-013-0522-6. Epub 2013 Oct 17. PMID 24132660
- [Derived] Bozzetto L, Prinster A, Annuzzi G, Costagliola L, Mangione A, Vitelli A, Mazzarella R, Longobardo M, Mancini M, Vigorito C, Riccardi G, Rivellese AA. Liver fat is reduced by an isoenergetic MUFA diet in a controlled randomized study in type 2 diabetic patients. Diabetes Care. 2012 Jul;35(7):1429-35. doi: 10.2337/dc12-0033. PMID 22723581